CLINICAL TRIAL: NCT01235130
Title: Phase 3 A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Effect of Long-chain N-3 Polyunsaturated Fatty Acids (OMEGA-3) on Arrhythmia Recurrence in Atrial Fibrillation
Brief Title: Multi_center Study to Evaluate the Effect of N-3 Fatty Acids (OMEGA-3) on Arrhythmia Recurrence in Atrial Fibrillation
Acronym: AFFORD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCT88068; MCT88068 (Other Grant/Funding Number: CIHR MCT88068)
Record Dates: First submitted 2010-07-29; First posted 2010-11-05 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OMEGA-3 (Active Comparator): Long-Chain N-3 polyunsaturated fatty acids (OMEGA-3)
  Interventions: Drug: OMEGA-3
- Placebo (Placebo Comparator): Placebo soybean oil
  Interventions: Drug: Placebo soybean oil

INTERVENTIONS:
Drug: OMEGA-3 — 600mg, 2 caps, twice a day
  Other Names: Long-chain N-3 polyunsaturated fatty acids
  Arms: OMEGA-3
Drug: Placebo soybean oil — 600mg, 2caps twice a day
  Arms: Placebo

SUMMARY:
The general objective of this study is to demonstrate the effectiveness of n-3 fatty acids, 2.4 grams per day, to prevent recurrence of atrial fibrillation in patients with paroxysmal or persistent AF in whom a rhythm-control strategy is planned.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) represents the most common arrhythmia of clinical importance. The prevalence of AF in the general population has been estimated to be just below 1%, or 300,000 Canadians, and rising. Current strategies in AF to preserve normal sinus rhythm include pharmacological therapy with agents that demonstrate intermediate efficacy and significant adverse effects. Newer non-pharmacological strategies such as pulmonary vein ablation are suitable for only a minority of patients and are an expensive method of treatment. As a result, simple, safe, inexpensive and effective strategies to treat AF and preserve sinus rhythm are required given the great health and financial burden that this condition represents to our society.

Omega-3 or "n-3" polyunsaturated fatty acids (n-3 fatty acids) represent a novel approach to the prevention and treatment of AF. N-3 fatty acids have known anti-arrhythmic properties and are associated with a lower risk of sudden (arrhythmic) death. Additionally, n-3 fatty acids have significant anti-inflammatory properties and potential anti-oxidant effects. Higher consumption of non-fried fish was recently shown to confer a lower incidence of new onset AF in elderly adults. N-3 fatty acids might therefore represent a useful strategy for maintenance of sinus rhythm in patients with AF, given their potential to act on several mechanisms simultaneously. We seek to test this hypothesis in the current clinical trial proposal.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Written informed consent
3. Non-valvular paroxysmal or persistent AF in whom a rhythm control strategy is planned
4. Duration of at least one symptomatic AF episode > 10 minutes within the past 6 months
5. ECG documentation of AF

Exclusion Criteria:

1. Chronic AF (continuously present for > 3 months)
2. Myocardial infarction within the past month prior to selection visit
3. Cardiac or thoracic surgery within the past 3 months or likely to be performed during trial
4. Moderate to severe congestive heart failure (NHYA FC III-IV)
5. Known left ventricular dysfunction (EF< 40%).
6. Mitral stenosis
7. Moderate to severe mitral insufficiency (Grade 3-4/4)
8. AF secondary to an acute reversible condition (untreated or uncontrolled hyperthyroidism, post- operative AF, fever, anemia)
9. Need for anti-arrhythmic therapy for a condition other than atrial fibrillation
10. Wolff-Parkinson-White syndrome
11. Any medical condition making compliance with study treatment unlikely
12. Current use of n-3 fatty acid supplements or use within the past 3 months
13. Pregnancy, breastfeeding, or possibility of becoming pregnant during the study (Patients must have adequate contraception as determined by the investigator),
14. Participation in another study at the same time or within 30 days of randomization.
15. Uncontrolled hypertension (systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg
16. Suspected or known allergy to any ingredients in the study product or placebo, fish or shellfish .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Time to first relapse of atrial fibrillation | After a three weeks loading phase
  The primary endpoint will be the time to first relapse of AF during the follow-up period. Relapse is defined as any ECG-documented episode of AF lasting longer than 30 seconds, symptomatic or asymptomatic. ECG-documented AF refers to episodes documented either by trans-telephonic event recorder, 12-lead ECG or Holter monitor.

SECONDARY OUTCOMES:
High Sensitivity C-Reactive protein level | Measured at 0 and 6 months
  Based upon the primary endpoint, to demonstrate a relative reduction in CRP levels between the 2 groups
Cardiovascular-related death or Hospitalisation | At each scheduled visit (3 weeks, 4 weeks, 7 weeks, 15 weeks, 27 weeks, 47 weeks and 67 weeks)
  Data on CV-related hospitalization will be collected prospectively during scheduled patient visits with patients being asked about any emergency room visits, hospital admissions or bleeding since their last scheduled visit.
Serum myeloperoxidase level | Measured at 0 and 6 months
  Based upon the primary endpoint, to demonstrate a relative reduction in MPO levels between the 2 groups
Major bleeding | At each scheduled visit (3 weeks, 4 weeks, 7 weeks, 15 weeks, 27 weeks, 47 weeks and 67 weeks)
  Data on bleeding episodes will be collected prospectively during scheduled patient visits with patients being asked about any emergency room visits, hospital admissions or bleeding since their last scheduled visit.
Quality of life data | Measured at 0 week, 27 weeks, 47 weeks, and 67 weeks
  Quality of life will be evaluated using questionnaires: Toronto Atrial Fibrillation Severity Scale (AFSS), Severity of Atrial Fibrillation Scale (SAF), SF-12, EuroQol-5, Anxiety Severity Scale and Beck Depression Inventory-II.
Resource utilization | At each scheduled visit (3 weeks, 4 weeks, 7 weeks, 15 weeks, 27 weeks, 47 weeks and 67 weeks)
  Resource utilisation including drugs, cardioversions attempts, hospitalization days, emergency department visits, outpatient physician visits and pacemaker and catheter-based procedures will be recorded and converted to costs according to the methods described by the National List of provincial Cost Heath Care: Canada 1997/8.
Dietary habits | Measured at 0 week, 27 weeks, 47 weeks, and 67 weeks
  Dietary habits will be evaluated using a standardized food frequency questionnaire (FFQ).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anil Nigam, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute Coordinating Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nigam A, Talajic M, Roy D, Nattel S, Lambert J, Nozza A, Jones P, Ramprasath VR, O'Hara G, Kopecky S, Brophy JM, Tardif JC; AFFORD Investigators. Fish oil for the reduction of atrial fibrillation recurrence, inflammation, and oxidative stress. J Am Coll Cardiol. 2014 Oct 7;64(14):1441-8. doi: 10.1016/j.jacc.2014.07.956. PMID 25277614